CLINICAL TRIAL: NCT07265557
Title: A Pilot Randomized Controlled Trial Comparing Two Post-Operative Pain Protocols at Discharge for Orthopaedic Patients: A Pilot Study
Brief Title: Two Post-Operative Pain Protocols at Discharge for Orthopaedic Patients
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: McMaster University (Other)
Responsible Party: Principal Investigator, Arun Aneja, MD, PhD, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2025P002285
Record Dates: First submitted 2025-10-14; First posted 2025-12-05 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Orthopaedic Related Pain (Musculoskeletal Pain); Opioid; Pain; Pilot Study
Keywords: Opioid; Pilot study; Musculoskeletal Pain
MeSH Terms: conditions — Musculoskeletal Pain; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Discharge pain medication prescription without opioids (Experimental): The treatment arm will receive standard non-opioid analgesia, with the specific medication (e.g., ibuprofen, paracetamol, ketorolac) determined by the treating physician.
  Interventions: Other: Discharge pain medication prescription
- Usual care discharge prescription (with opioids) (Active Comparator): The control arm will receive the standard pain medication prescription, including opioids. The specific dosage and medication is determined by the treating physician.
  Interventions: Other: Discharge pain medication prescription

INTERVENTIONS:
Other: Discharge pain medication prescription — The patients in this pilot RCT will either receive a discharge prescription with or without opioids. The specific non-opioid medication (e.g., ibuprofen, paracetamol, ketorolac) determined by the treating physician. The dosage of the prescription including opioids is also determined by the treating physician.

SUMMARY:
This is a single-center, pilot randomized controlled trial designed to evaluate the feasibility of a definitive trial comparing opioid-free discharge prescriptions to usual care (which includes opioids) in patients undergoing major orthopaedic surgery. The main objective is to inform the design and feasibility of the definitive RCT.

DETAILED DESCRIPTION:
This is a single-center pilot RCT of at least 100 participants (20 participants from each subspecialty including trauma, arthroplasty, foot and ankle, spine, and sports) who undergo major orthopaedic surgery. Eligible and consenting patients will be randomized to either a discharge pain medication prescription without opioids or a usual care discharge pain medication (with opioids). The overarching objective of the pilot study is to inform the design and feasibility of the definitive RCT. For this pilot trial the investigators will measure feasibility against traffic light criteria based on enrollment metrics, treatment allocation adherence, and on data collection. Furthermore, this pilot RCT will compare the effectiveness of discharge pain medication without opioids to usual care discharge pain medication (with opioids) on opioid use and pain interference for patients who have undergone major orthopaedic surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older
2. Underwent a major operative orthopaedic procedure

Exclusion Criteria:

1. Contraindication for NSAIDs.
2. Preoperative chronic opioid use (preoperative use of >14 days and average of >30 Morphine Milligram Equivalents per day).
3. Active treatment for opioid use disorder.
4. Previous or current illicit drug use.
5. Major surgery for pathologic (cancer-related) condition.
6. Hand surgery.
7. Concurrent operative treatment by another specialty team.
8. Discharged to an extended medical care facility.
9. Incarceration.
10. Women who are pregnant or planning to become pregnant in the next 6 weeks.
11. Expected injury survival of less than 6 weeks.
12. Terminal illness with expected survival of less than 6 weeks.
13. Anticipated problems, in the judgment of research personnel, with maintaining follow-up with the patient.
14. Currently enrolled in a trial that does not permit co-enrollment.
15. Prior enrollment in the trial.
16. Unable to obtain informed consent.
17. Non-English speaking
18. Eligible patient was not approached prior to hospital discharge (missed participant).
19. Did not provide informed consent (declined participation).
20. Other reason to exclude the patient, as approved by the Principal Investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility of patient enrollment and treatment allocation | From enrollment to the end of the follow-up phase at 6 weeks
  Participant enrollment will be assessed by monitoring screening and enrollment metrics, including:
  * Participant enrollment
  * Feasibility of treatment allocation
  * Data collection methods (Proportion of participants with missing data)
  * Compliance with the protocol (Proportion of randomization errors, proportion of patients who complete each questionnaire at each of the follow-up, proportion of patients who withdraw from the trial, proportion of participants who are lost to follow-up)

SECONDARY OUTCOMES:
Opioid Use | From enrollment to the end of the follow-up at 6 weeks
  Opioid usage assessed at 2 weeks and 6 weeks post-randomization
Pain Interference | From enrollment to the end of the follow-up at 6 weeks
  Pain interference will be assessed using the Brief Pain Inventory at 2 weeks and 6 weeks from randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Arun Aneja, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Mass, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No